CLINICAL TRIAL: NCT06317337
Title: Effect of Focused Ultrasound Cavitation Augmented With Aerobic Exercise in Patients With Central Obesity
Brief Title: Focused Ultrasound Cavitation Augmented With Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sana Bshir
Record Dates: First submitted 2024-01-18; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Central Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- focused ultrasound cavitation augmented with aerobic exercise (Experimental): Ultrasound cavitation single session per week along with the Aerobic exercises. Aerobic Exercise was Treadmill walk for 30 min with moderate intensity
  Interventions: Other: focused ultrasound cavitation augmented with aerobic exercises
- focused ultrasound cavitation (Active Comparator): Ultrasound cavitation single session per week along with 6min walk test.
  Interventions: Other: focused ultrasound cavitation augmented with aerobic exercises

INTERVENTIONS:
Other: focused ultrasound cavitation augmented with aerobic exercises — Ultrasound cavitation single session per week along with the Aerobic exercises. Aerobic Exercise was Treadmill walk for 30 min with moderate intensity

SUMMARY:
This study will determine the combine effects of focused ultrasound cavitation augmented with aerobic exercises. This research could be helpful for the patients who prefer such treatments to make a wise decision that either aerobic exercises in combination with cavitation is the better and much safer treatment option to maintain healthy life.

DETAILED DESCRIPTION:
Abdominal obesity can be treated through invasive and non-invasive procedures. The most common invasive protocol is surgical liposuction, this is mostly useful for removing large volume of fat. Nonsurgical approaches included exercises and selective focus energy which target the subcutaneous adipose tissue including focused ultrasound. Focus ultrasound produce cavitation which results in fat cell lysis through mechanical energy without causing any harmful effect on surrounding nerves and connective tissue.

There is an increasing demand for noninvasive fat reduction methods; there is variety of physical treatments in practice for localized fat reduction such as electrical stimulation, mechanical massage, light based therapies and cold low level laser irradiation but clinically most of them failed to meet expectations. Literature reported that clinically High Intensity Focused Ultrasound (HIFU) is most effective for noninvasive fat reduction therapy. Ultrasound causes cavitation phenomena on fat droplet watery cytoplasm interface and eventually rupture of adipocytes and triglycerides release, this whole phenomena is caused through generation of compression and decompression cycle at specific frequency. Ultrasound Fat cavitation is the technique of handling obesity, specially by destroying fat and shaping a body part. There is a limited literature available on effects of aerobic exercises and focused ultrasound cavitation on obesity but there was no literature available on combine effects of both treatments. This study will determine the combine effects of focused ultrasound cavitation augmented with aerobic exercises. This research could be helpful for the patients who prefer such treatments to make a wise decision that either aerobic exercises in combination with cavitation is the better and much safer treatment option to maintain healthy life.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Overweight (Asian BMI scoring)
* 25 to 40 years of age
* Central obesity

Exclusion Criteria:

* Morbidly obesity
* Hypertension
* Arthritis
* Musculoskeletal disorders
* Cardiovascular disorders

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female with central obesity
Enrollment: 54 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Borg rating of perceived exertion scale | 4 weeks
  The Borg Rating of Perceived Exertion (RPE) scale, developed by Swedish researcher Gunnar Borg, is a tool for measuring an individual's effort and exertion, breathlessness and fatigue during physical work and so is highly relevant for occupational health and safety practice. In its simplest terms, it provides a measure of how hard it feels that the body is working based on the physical sensations that the subject experiences, including increased heart rate, increased respiration or breathing rate, increased sweating and muscle fatigue.
girth | 4weeks
  Anthropometry is the measurement of human body dimension such as girths by using surface landmarks for reference. Like other areas of science the procedures and processes depend upon adherence to the particular rules of measurement as determined by national and international standards bodies. The definitions and instructions in this chapter are consistent with the international anthropometric standards body called the International Society for the Advancement of Kinanthropometry (ISAK).
6min walk test | 4weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity

CONTACTS AND LOCATIONS:
Overall Officials: Maria Razzaq, MSCPPT, Principal Investigator — Riphah International university Gulberg Greens D block Islamabad
Locations (1):
- Bioflex Aesthetic Clinic, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No